CLINICAL TRIAL: NCT01607099
Title: Sodium Picosulfate Plus Magnesium Citrate Versus Macrogol 4000 in the Bowel Cleansing Procedure: a Comparison of Efficiency and Compatibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PicoPrep
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Laxative Compatibility
Keywords: colonoscopy; bowel cleansing; bowel cleanness; efficiency; compatibility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pico Prep (Experimental): Arm in which sodium- picosulfate/magnesium citrate is used for bowel cleansing
  Interventions: Procedure: Compatibility
- Standard (No Intervention): The standard drug macrogol is used for bowel cleansing

INTERVENTIONS:
Procedure: Compatibility — Patients asses the compatibility of the bowel cleansing procedure
  Arms: Pico Prep

SUMMARY:
For effective cleansing of the bowel prior to colonoscopy polyethylene glycol (e.g. macrogol) has widely been used in Germany. Usually patients have to drink between 4 an 6 liter of macrogol in a split dose (3 liter on the day before and 1 to 3 liter on the of the examination). One handicap of using polyethylene glycol is the occurence of nausea and vomiting which is due to the high amount of the laxativ and its bad taste. Therefore in a pilot study the investigators have detected a high fraction of patients who consider the cleansing procedure wich macrogol as "very distressing". Thus patient acceptance of the colonoscopy procedure altogether is low.

Since a few month sodium picosulfate/magnesium citrate is available for bowel cleansing in Germany. This preparation tastes better and needs less fluid intake. Usually 150 ml of sodium picosulfate/magnesium citrate are given twice within a 12 hour interval. Patients are instructed to drink plenty of water in addition to the laxative. In the mentioned pilot study the investigators found the cleansing procedure with picosulfate/magnesium citrate to be much more compatible compared to the macrogol regime. The effectiveness expressed by the cleanness of the bowel was equal in both groups.

The investigators believe that a new protocol which contains sodium picosulfate/magnesium citrate instead of macrogol will benefit the patients by fewer abdominal side effects while cleanness of the bowel at the same time will be warranted. This presumption is the reason for the present study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Scheduled for colonoscopy

Exclusion Criteria:

* No informed consent
* ASA IV or V
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-09; Primary Completion 2014-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Valuation "very distressing" | Just before colonoscopy up to 4 hours afterwards (0 to aprox 4 hours)
  Patients will fill in a report in which they rate the stress triggered by the bowel cleansing procedure. The level ranges from 1 to 10 points. Valuations from 8 to 10 points will be considered as very distressing.

SECONDARY OUTCOMES:
Colon cleanness | From the start to the end of colonoscopy, i.e. from 0 h to approximately 2 h

CONTACTS AND LOCATIONS:
Overall Officials: Peter Klare, MD, Principal Investigator — Technical University of Munich; Wolfgang Huber, MD, Study Director — Technical University of Munich
Locations (1):
- Technische Universität München, Munich, Bavaria, Germany